CLINICAL TRIAL: NCT02746640
Title: Prospective Assessment Project About Cardiac Arrest Resuscitation
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: PAPA CARES
Record Dates: First submitted 2016-04-05; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiopulmonary resuscitation (CPR) — If there is a cardiopulmonary arrest, investigators observe the working processes of cardiopulmonary resuscitation.

SUMMARY:
In case of a cardiac arrest it is very important to quickly provide high quality cardiopulmonary resuscitation (CPR). For reasons of patient safety the investigators want to assess the frequency, the quality and the outcome of cardiopulmonary resuscitations in the Inselspital Bern.

ELIGIBILITY:
Inclusion Criteria:

* Every patient for which the alarm button for a cardiopulmonary arrest gets triggered

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient, for which the alarm button for a cardiopulmonary arrest gets triggered will be included and observate.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of reanimation alarms during a time period of 1 year. | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuchs A, Kaser D, Theiler L, Greif R, Knapp J, Berger-Estilita J. Survival and long-term outcomes following in-hospital cardiac arrest in a Swiss university hospital: a prospective observational study. Scand J Trauma Resusc Emerg Med. 2021 Aug 11;29(1):115. doi: 10.1186/s13049-021-00931-0. PMID 34380539